CLINICAL TRIAL: NCT02384798
Title: Noninvasive Ventilatory Support Associated With Concurrent Training in Improved Functional Capacity and Quality of Life in Patients With Heart Failure
Brief Title: Ventilatory Support Associated With Exercise in Heart Failure
Acronym: SVNI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Collaborators: Hospital Ana Nery (Other)
Responsible Party: Principal Investigator, Mansueto Gomes Neto, Physiotherapy course coordinator, Federal University of Bahia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FUBahia914311
Record Dates: First submitted 2015-02-16; First posted 2015-03-10 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ventilatory support (Experimental): noninvasive ventilatory support to 5cmH2O used before the session of interval training and resistance exercises performed three times a week for 12 weeks
  Interventions: Other: noninvasive ventilatory support; Other: interval training
- interval training (Active Comparator): sessions of interval training and resistance exercises performed three times a week for 12 weeks
  Interventions: Other: interval training

INTERVENTIONS:
Other: noninvasive ventilatory support — noninvasive ventilatory support with 5-minute ramp and positive end expiratory pressure (PEEP) of 5 cm H2O for 30 minutes, then there will be the interval aerobic training on a treadmill added to resistance exercises
  Other Names: CPAP of redmed brand
  Arms: ventilatory support
Other: interval training — interval training
  Other Names: concurrent training

SUMMARY:
Due to the symptoms of heart failure (HF), as dyspnea and fatigue, patients have a reduced functional capacity, evidenced during usual daily activities and exercises. The Cardiac Rehabilitation with emphasis on resistance and aerobic exercises performed in the same session (concurrent training), can be added to pharmacological treatment as improvement strategy in functional capacity and quality of life.

DETAILED DESCRIPTION:
A randomized clinical trial, divided into two stages will be held. In step 1 the function will be assessed by the 6-minute walk test, spirometry, and questionnaires to evaluate quality of life. After fulfilled the series of assessments individuals will be randomly divided into two groups, with group 1 (control) will hold only one interval aerobic exercise program on treadmill and group 2 (intervention) will hold a combined exercise program for prior use of ventilatory support noninvasive. For both groups will be held an aerobic exercise program associated with resistance exercise for 12 weeks. The first two weeks will be considered in period. In the 10 weeks following both groups maintain the preset exercise program gradually. In the intervention group will be added before the exercise program the use of noninvasive ventilation for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Will be included 60 patients of both sexes, adults with medical diagnosis divided into two groups: Group A consisted of 30 patients use non-invasive ventilation added to interval training and group B consisted of 30 patients also only use interval training.

Exclusion Criteria:

* Will be excluded from the study patients who have chest pain (angina), arrhythmias, spo2 ≤ 90%, hypertension or hypotension, neurological or osteoarticular disease preventing the ambulation of these individuals.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
SIX MINUTES WALK TEST | AFTER 12 WEEKS FOLLOW
  Identifying whether a combined resistance and aerobic exercise program (concurrent training) associated with the use of non-invasive ventilation is effective in improving the quality of life and functional capacity of patients with ventricular dysfunction.

SECONDARY OUTCOMES:
double product | AFTER 12 WEEKS FOLLOW
  Identifying whether a combined resistance and aerobic exercise program (concurrent training) associated with the use of non-invasive ventilation is effective in improving the quality of life and functional capacity of patients with ventricular dysfunction.
spirometry | AFTER 12 WEEKS FOLLOW
  Identifying whether a combined resistance and aerobic exercise program (concurrent training) associated with the use of non-invasive ventilation is effective in improving the quality of life and functional capacity of patients with ventricular dysfunction.
minnesota questionnaire | AFTER 12 WEEKS FOLLOW
  Identifying whether a combined resistance and aerobic exercise program (concurrent training) associated with the use of non-invasive ventilation is effective in improving the quality of life and functional capacity of patients with ventricular dysfunction.
SF-36 questionnaire | AFTER 12 WEEKS FOLLOW
  Identifying whether a combined resistance and aerobic exercise program (concurrent training) associated with the use of non-invasive ventilation is effective in improving the quality of life and functional capacity of patients with ventricular dysfunction.
Functional Independence Measure questionnaire | AFTER 12 WEEKS FOLLOW
  Identifying whether a combined resistance and aerobic exercise program (concurrent training) associated with the use of non-invasive ventilation is effective in improving the quality of life and functional capacity of patients with ventricular dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: MANSUETO G NETO, Principal Investigator — Federal University of Bahia

REFERENCES:
- [Result] Paterson JM, Smith SM, Simpson J, Grace OC, Sosunov AA, Bell JE, Antoni FA. Characterisation of human adenylyl cyclase IX reveals inhibition by Ca(2+)/Calcineurin and differential mRNA plyadenylation. J Neurochem. 2000 Oct;75(4):1358-67. doi: 10.1046/j.1471-4159.2000.0751358.x. PMID 10987815
- [Derived] Bittencourt HS, Cruz CG, David BC, Rodrigues E Jr, Abade CM, Junior RA, Carvalho VO, Dos Reis FBF, Gomes Neto M. Addition of non-invasive ventilatory support to combined aerobic and resistance training improves dyspnea and quality of life in heart failure patients: a randomized controlled trial. Clin Rehabil. 2017 Nov;31(11):1508-1515. doi: 10.1177/0269215517704269. Epub 2017 Apr 5. PMID 28378600